CLINICAL TRIAL: NCT03593564
Title: Knowledge and Interpersonal Skills to Develop Exemplary Relationships
Acronym: KINDER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team experienced technology challenges with the digital platform used to deliver the intervention and to collect data. Data collection surveys would be automatically sent to participants before participants completed intervention modules.
Sponsor: University of Southern California (Other)
Collaborators: Archstone Foundation (Other)
Responsible Party: Principal Investigator, Donna Benton, Research Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KINDER 18-01-06
Record Dates: First submitted 2018-06-26; First posted 2018-07-20 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Caregivers; Family Relations; Domestic Violence; Elder Abuse
Keywords: Pilot Study; Cognitive Behavioral Therapy; Intervention Study

STUDY DESIGN:
Intervention Model Description: The investigators will evaluate the KINDER program using pre- and post-test analysis. Eligible and consented subjects enrolled on a rolling basis. After enrollment, all caregivers will complete a baseline assessment. Caregivers will receive the intervention (8 lessons, delivered once per week) and will be asked to complete a reassessment after 10 weeks. Two months later, participants will be asked to complete a second reassessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KINDER Participant (Experimental): The intervention will be provided with a 8-part psychoeducational intervention delivered online on a weekly basis. Online modules will be comprised of a short (approximately 3 minute) videos followed by more specific text-based information and links to additional resources. At the end of the module, participants will complete a short quiz, followed by a reflection exercise to reinforce learning. Each model, participants will be asked to select a goal to complete a pleasurable activity and receive an option to set a text or email reminder to do so.
  Interventions: Behavioral: KINDER

INTERVENTIONS:
Behavioral: KINDER — KINDER is an online course for people assisting an older adult with dementia. It is intended to improve the quality of caregiver's relationship with the care recipient and reduce the chance of risky relationship behavior (e.g., yelling). Courses will cover topics including understanding cognitive impairments, navigating evolving roles, and dealing with frustration. During this course, participants will learn skills to deal with difficult situations caregivers frequently encounter in ways that support a healthy caregiving relationship. Videos will be story-based and represent different types of caregiving relationships and challenges encountered.

SUMMARY:
This pilot study will test the effect of an online asynchronous psychoeducational intervention to improve relationship quality and prevent verbal-type elder mistreatment in caregiving dyads. The investigators will use a pre-post test design to test the feasibility and acceptability of this video-based intervention, and to determine the likelihood that participation in this program may improve caregiver relationship quality.

ELIGIBILITY:
Inclusion Criteria:

* Provides assistance to someone over the age of 60 with an illness or a disability ("care recipient") who requires personal assistance from another person (e.g., bathing, preparing meals). (Assistance provided with at least 1 activity of daily living and/or at least 2 instrumental activities of daily living.)
* Person receiving care from the study participant has a cognitive impairment. This does not have to be diagnosed.
* Participant provides at least 8 hours of assistance to the care recipient per week
* Participant does not intend to place the care recipient in a skilled nursing facility or assisted living facility within 3 months of consenting into the study

Exclusion Criteria:

* Does not read and speak English
* Cannot access a computer and internet (needed to complete lessons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Change in frequency of verbal mistreatment | This measure will be asked immediately before the intervention, immediately after the intervention, and 2 months after the intervention is complete. The question asks participants about events in the previous 2 months.
  This scale will measure frequency of verbal mistreatment using a measure based on the Conflict Tactics Scale (Straus et al., 1996), with additional questions from other items (Acierno et al., 2010; Beach et al., 2005; Conrad et al., 2011; Deliema et al., 2012)
Change in the number of positive aspects of the relationship with the care recipient (Dyadic Relationship Scale) | This measure will be asked immediately before the intervention, immediately after the intervention, and 2 months after the intervention is complete. The question asks participants about events in the previous 2 months.
  Participants are asked how much they agree with positive statements about their relationship with the care receiver on a 0 to 3 scale. This item comes from Sebern & Whitlatch (2007)

SECONDARY OUTCOMES:
Change in caregiver competence (Caregiving Competence Scale) | This measure will be asked immediately before the intervention, immediately after the intervention, and 3 months after the intervention is complete. The question asks participants about events in the previous 3 months.
  We will use the Caregiving Competence Scale developed by Pearlin and colleagues (1990)
Change in perceived stress (Perceived Stress Scale) | This measure will be asked immediately before the intervention, immediately after the intervention, and 3 months after the intervention is complete. The question asks participants about events in the previous 3 months.
  We will use the Perceived Stress Scale developed by Cohen & Williamson (1988)
Change in caregiver burden (Zarit Burden Index) | This measure will be asked immediately before the intervention, immediately after the intervention, and 3 months after the intervention is complete. The question asks participants about events in the previous 3 months.
  We will use the Zarit Burden Index developed by Zarit and colleagues (1980)
Change in depression (Patient Health Questionnaire-9) | This measure will be asked immediately before the intervention, immediately after the intervention, and 3 months after the intervention is complete. The question asks participants about events in the previous 3 months.
  We will use the Patient Health Questionnaire-9 (Kroenke et al., 2001)
Change in caregiver mastery (Caregiver Mastery Scale) | This measure will be asked immediately before the intervention, immediately after the intervention, and 3 months after the intervention is complete. The question asks participants about events in the previous 3 months.
  We will use the Caregiver Mastery Scale developed by Pearlin & Schooler (1978)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Benton, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified participant data will be available to other researchers at the end of our study.

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Straus, M. A., Hamby, S. L., Boney-McCoy, S., Sugarman, D. B. The revised conflict tactics scales (CTS2) development and preliminary psychometric data. Journal of Family Issues 17(3): 283-316, 1996.
- [Background] DeLiema M, Gassoumis ZD, Homeier DC, Wilber KH. Determining prevalence and correlates of elder abuse using promotores: low-income immigrant Latinos report high rates of abuse and neglect. J Am Geriatr Soc. 2012 Jul;60(7):1333-9. doi: 10.1111/j.1532-5415.2012.04025.x. Epub 2012 Jun 14. PMID 22697790
- [Background] Acierno R, Hernandez MA, Amstadter AB, Resnick HS, Steve K, Muzzy W, Kilpatrick DG. Prevalence and correlates of emotional, physical, sexual, and financial abuse and potential neglect in the United States: the National Elder Mistreatment Study. Am J Public Health. 2010 Feb;100(2):292-7. doi: 10.2105/AJPH.2009.163089. Epub 2009 Dec 17. PMID 20019303
- [Background] Conrad KJ, Iris M, Ridings JW, Langley K, Anetzberger GJ. Self-report measure of psychological abuse of older adults. Gerontologist. 2011 Jun;51(3):354-66. doi: 10.1093/geront/gnq103. Epub 2010 Dec 20. PMID 21173437
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Pearlin LI, Schooler C. The structure of coping. J Health Soc Behav. 1978 Mar;19(1):2-21. No abstract available. PMID 649936
- [Background] Cohen, S, Williamson, G. Perceived stress in a probability sample of the United States. In S. Spacapan & S. Oskamp (Eds.), The social psychology of health: Claremont Symposium on applied social psychology. Newbury Park, CA: Sage, 1988
- [Background] Pearlin LI, Mullan JT, Semple SJ, Skaff MM. Caregiving and the stress process: an overview of concepts and their measures. Gerontologist. 1990 Oct;30(5):583-94. doi: 10.1093/geront/30.5.583. PMID 2276631
- [Background] Beach SR, Schulz R, Williamson GM, Miller LS, Weiner MF, Lance CE. Risk factors for potentially harmful informal caregiver behavior. J Am Geriatr Soc. 2005 Feb;53(2):255-61. doi: 10.1111/j.1532-5415.2005.53111.x. PMID 15673349
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628